CLINICAL TRIAL: NCT02803177
Title: BMC2012, Cell Based Therapy by Implanted Bone Marrow-derived Mononuclear Cells (BMC) for Bone Augmentation of Plate-stabilized Proximal Humeral Fractures - a Randomized, Open, Multicentric Study - Phase IIa
Brief Title: Cell Therapy by Autologous BMC for Large Bone Defect Repair
Acronym: BMC2012
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: LOEWE CGT (Unknown)
Responsible Party: Principal Investigator, Ingo Marzi, MD Prof., head physician, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMC2012 Phase IIa
Record Dates: First submitted 2016-06-07; First posted 2016-06-16 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Humerus Fracture Displaced Proximal
Keywords: large bone defect; bone marrow-derived mononuclear cells

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMC2012 + beta-TCP Chronos® Synthes (Experimental): The large bone defect will be bridged as per clinical standard, filled with a clinically established scaffold (beta-TCP Chronos® Synthes), and loaded with 1.3 x 10E6 BMC/ml TCP per 1 ml beta-TCP in situ.
  Interventions: Biological: BMC2012
- beta-TCP Chronos® Synthes (Placebo Comparator): The large bone defect will be bridged as per clinical Standard and filled with a clinically established scaffold (beta-TCP Chronos® Synthes).
  Interventions: Device: beta-TCP Chronos® Synthes

INTERVENTIONS:
Biological: BMC2012
  Arms: BMC2012 + beta-TCP Chronos® Synthes
Device: beta-TCP Chronos® Synthes
  Arms: beta-TCP Chronos® Synthes

SUMMARY:
In the present phase-II clinical trial the researchers investigate efficacy and proof of concept of the augmentation with preoperatively isolated autologous BMC cells seeded onto ß-TCP in combination with an angle stable fixation (Philos plate®) for the therapy of proximal humeral fractures.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 50. and 90. years with proximal humerus fractures
* indication for open reposition and internal stabilisation with a proximal fixed- angle plate for humerus (PHILOS, Synthes, Oberdorf, Swiss):
* 2-, 3- or 4-fragment fracture according to Neer
* dislocation of >10 mm between fragments and/or
* angle of > 45° between fragments and/or
* dislocation of tuberculum majus > 5 mm
* negative pregnancy test of premenopausal women
* signed informed consent for surgery and participation in the clinical trial

Exclusion Criteria:

* contraindications against administration of Investigational medicinal product (IMP) is pregnancy and nursing
* dislocation fracture
* known psychic disorder that leads to incompliance (e.g. dementia, schizophrenia, major depression)
* pathologic fractures caused by other underlying diseases
* fracture-induced nerve damage
* tumor disease with recent adjuvant therapy or treatment during the last 3 months (e.g. chemotherapy, radiotherapy), untreated tumor diseases
* known hypersensibility against components of the transplant
* participation in a clinical trial during the last 3 months prior to this study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Secondary dislocation of fracture | 12 weeks
  Secondary dislocation is diagnosed on plain radiographs, if more than 20° varus collapse of the humeral head fragment in relation to the humeral shaft and / or screw penetration through the humeral head is detected

SECONDARY OUTCOMES:
Functional outcome after fixation | 12 weeks
  Functional outcome after fixation will be recorded by the Dash-Score at week 12; assessment of safety: all adverse reactions will be recorded and analyzed.

OTHER OUTCOMES:
Concomitant medication | day -1
  Documentation of concomitant medication
Adverse events | day -1
  Documentation of adverse events
Concomitant medication | day 0
  Documentation of concomitant medication
Adverse events | day 0
  Documentation of adverse events
Concomitant medication | week 1
  Documentation of concomitant medication
Adverse events | week 1
  Documentation of adverse events
Concomitant medication | week 6
  Documentation of concomitant medication
Adverse events | week 6
  Documentation of adverse events
Concomitant medication | week 12
  Documentation of concomitant medication
Adverse events | week 12
  Documentation of adverse events
Degree of bony bridging (percent of defect area) in the bone fracture | week 1
  Analysis of fracture healing by radiologic evaluation, consolidation, necrosis
Degree of bony bridging (percent of defect area) in the bone fracture | week 6
  Analysis of fracture healing by radiologic evaluation, consolidation, necrosis
Degree of bony bridging (percent of defect area) in the bone fracture | week 12
  Analysis of fracture healing by radiologic evaluation, consolidation, necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Marzi, MD Prof., Principal Investigator — Department of Trauma-, hand- and reconstructive surgery, Goethe University, Frankfurt
Locations (1):
- Department of trauma-, hand- and reconstructive surgery, Goethe University, Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
The researchers will only publish data in their scientific publication

REFERENCES:
- [Derived] Seebach C, Nau C, Henrich D, Verboket R, Bellen M, Frischknecht N, Moeck V, Eichler K, Horlohe KHS, Hoffmann R, Bonig H, Seifried E, Frank J, Marzi I. Cell-Based Therapy by Autologous Bone Marrow-Derived Mononuclear Cells for Bone Augmentation of Plate-Stabilized Proximal Humeral Fractures: A Multicentric, Randomized, Open Phase IIa study. Stem Cells Transl Med. 2024 Jan 12;13(1):3-13. doi: 10.1093/stcltm/szad067. PMID 37995325